CLINICAL TRIAL: NCT00116870
Title: A Double-Blind, Placebo-Controlled Angiographic Study to Evaluate the Effect of Lovastatin on the Progression Rate of Atherosclerosis in the Coronary Arteries of Patients With Coronary Heart Disease
Brief Title: MARS - Monitored Atherosclerosis Regression Study
Status: Completed | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Organization: National Institute on Aging (NIA) (NIH)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: AG0027; MK-803
Record Dates: First submitted 2005-06-30; First posted 2005-07-01 (Estimated); Last update posted 2009-12-11 (Estimated); Status verified 2005-06

CONDITIONS: Atherosclerosis; Coronary Artery Disease
Keywords: CAD; familial hypercholesterolemia
MeSH Terms: conditions — Atherosclerosis; Coronary Artery Disease; Hyperlipoproteinemia Type II | interventions — Lovastatin

INTERVENTIONS:
Drug: lovastatin

SUMMARY:
The purpose of this study is to determine whether significant alterations in serum lipoproteins as provided by the drug lovastatin can substantially reduce atherosclerosis progression or even induce regression.

DETAILED DESCRIPTION:
Two conceptual advances occurring in the 1980's made it possible to test the hypothesis that significant alterations in serum lipoproteins can substantially reduce atherosclerosis progression or even induce regression. The first advance was in the development of arteriograms used in characterizing atherosclerosis, greatly reducing the number of patients required for the evaluation of an intervention designed to prevent coronary atherosclerosis progression. The second advance was the development of lovastatin that provides a lipid-lowering alternative much easier to tolerate than the niacin/colestipol combination previously used, and has been shown to be comparably effective for LDL reduction in patients with a family history of high cholesterol.

A total of 270 high-risk coronary artery disease patients, not eligible for coronary artery bypass surgery, were recruited for the study. All patients received angiograms and were randomly assigned to either the lovastatin or placebo groups stratified by three baseline factors: sex, smoking status, and plasma cholesterol levels.

Patients initially received lovastatin 40mg twice a day or a matching placebo. Those patients receiving lovastatin whose total plasma cholesterol level was less than 110mg/dL at one visit or 120 mg/dL on two successive visits had their dosage halved, and were maintained on the optimal dosage for the remainder of the study. Coronary angiography was performed prior to screening and at month 24 (visit 18). Angiographic assessment of both femoral arteries was also performed at baseline and at month 24. Noninvasive ultrasound imaging of the carotid arteries (including carotid intima-media thickness) was performed every 6 months. Patients reported to the clinic monthly for 12 months, and at two-month intervals thereafter. Plasma lipids, routine laboratory safety and physical examinations were also performed.

ELIGIBILITY:
Inclusion Criteria:

* Angiography within 17 weeks of randomization showing patient is at high risk for coronary artery disease but not a candidate for coronary artery graft surgery
* Men and women ages 21 through 67 years
* Mean plasma cholesterol levels from the first two screening visits in the range of 190 to 270 mg/dL
* Smokers are admitted, but encouraged to stop smoking tobacco

Exclusion Criteria:

* Premenopausal women unless surgically sterilized
* Hypertension, diabetes, thyroid disease, liver dysfunction, renal insufficiency, congestive heart failure, major arrhythmia, left ventricular conduction defects
* Physical impairment that may interfere with participation
* Life threatening disease with high likelihood of disability or death during the trial period
* Use of hydralazine, guanethidine, lipid-lowering drugs, estrogens, steroids, amphetamines, antibiotics, theophylline, acetaminophen (average daily use greater than ten grains), other drugs as determined by the principle investigator
* Vitamins A or D in doses greater than the Recommended Daily Allowance (RDA)
* Alcohol abuse
* Nutritional supplements high in cholesterol content
* Chelation therapy
* Psychosocial situations which make completion of the study unlikely
* Hypersensitivity to any component of the study medication

Ages: 21 Years to 67 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 1985-06; Primary Completion 1992-02 (Actual); Study Completion 1992-02 (Actual)

PRIMARY OUTCOMES:
the average (per-patient) change from baseline in percent diameter stenosis in all lesions that showed 20% diameter stenosis at baseline or at follow-up as evaluated by quantitative coronary angiography

SECONDARY OUTCOMES:
average (per-patient) change in minimum lumen diameter assessed by quantitative angiography
the global change score assessed by a human panel
the proportion of patients with progression or regression of disease assessed by quantitative coronary angiography

CONTACTS AND LOCATIONS:
Overall Officials: Howard N. Hodis, MD, Principal Investigator — University of Southern California, Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine
Locations (1):
- Atherosclerosis Research Unit, Division of Cardiovascular Medicine, Department of Medicine, Los Angeles, California, United States